CLINICAL TRIAL: NCT06861231
Title: Combined Intervention Using Transcranial Direct Current Stimulation and Cognitive Training in Alzheimer's Type Dementia Patients
Brief Title: Combined tDCS and Cognitive Training in Alzheimer's
Acronym: COMBINA-COG
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan Carlos Melendez, Professor of Psychology, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2601758
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Prodromal Alzheimer's Disease
Keywords: Cognitive impairment; Transcranial direct current stimulation; Cognitive training
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS active and cognitive training (Experimental): tDCS: HDC stimulator will be used. For active stimulation, it will be programmed with a constant current intensity of 2mA and a stimulation time of 20 minutes daily for 12 days, with an initial and final ramp of 30 seconds. A neoprene cap based on the international 10-10 EEG system will be used for current passage to the skull. The electrodes will have two sponges (5 x 5 cm) soaked in saline solution for contact with the skull. The anode will be placed over the left dorsolateral prefrontal cortex (DLPFC), and the cathode will be placed over the right supraorbital area (rSO).
  Cognitive training consists of a total of 12 sessions lasting 50 minutes each. These sessions will primarily focus on tasks involving executive functions and memory for a similar duration in each session. At the beginning of the sessions, instructions will be explained, followed by handing out activity sheets. The emphasis will not be on the outcome but on the cognitive activation process.
  Interventions: Device: Transcraneal Direct Current Stimulation (tDCS)- Active; Behavioral: Cognitive Training (CT)
- tDCS sham and cognitive training (Active Comparator): For the active comparator group, the stimulator will be programmed so that patients will receive direct current only during the ramps to generate the sensation of the current. Thus, it will enter a current pause after completing the initial ramp and will be activated in the final seconds during the final ramp. The cognitive training program will have the same characteristics as in the experimental group.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)- Sham; Behavioral: Cognitive Training (CT)

INTERVENTIONS:
Device: Transcraneal Direct Current Stimulation (tDCS)- Active — The stimulation will use a neoprene cap with carbon rubber electrodes and sponges soaked in saline solution (5x5 cm). The anode will be placed over the left dorsolateral prefrontal cortex (DLPFC), and the cathode over the right supraorbital area (rSO). Constant current intensity of 2mA and a stimulation time of 20 minutes per day for 12 days will be applied, with an initial and final ramp of 30 seconds.
  Arms: tDCS active and cognitive training
Device: Transcranial Direct Current Stimulation (tDCS)- Sham — Participants assigned to the sham tDCS group will also receive 12 home-based sessions of 20 minutes each. However, to mimic the sensation of active stimulation without delivering therapeutic current, the stimulator will only apply current during the initial and final 30-second ramp periods. The device will remain on for 20 minutes, but no current will be applied after the first ramp, simulating an active procedure without physiological effect.
  Arms: tDCS sham and cognitive training
Behavioral: Cognitive Training (CT) — All participants will complete 12 home-based cognitive training sessions, each lasting 50 minutes. The training will include structured tasks focused on executive function and memory, such as categorization, problem-solving, autobiographical recall, planning, and schedule analysis. Instructions will be provided at the start of each session, and participants will work independently or with caregiver support.

SUMMARY:
The General Objective of the study is to evaluate the short- and long-term efficacy of combining transcranial Direct Current Stimulation (tDCS) and cognitive training (CT) in patients with mild cognitive impairment and early-stage Alzheimer's disease. A randomized, double-blind, placebo-controlled design will be applied. An inter-subject design with two groups will be used: a. Active tDCS + concurrent CT and b. Sham tDCS + concurrent CT. Evaluations will be taken at pre-test, post-test, and follow-up one month later. The hypothesis comparing active and sham tDCS with concurrent CT is that, although both groups should improve due to concurrent CT, it is expected that the active tDCS group will show significantly greater improvements in post-treatment. Additionally, these improvements should be maintained in the long-term follow-up in the active tDCS group, while in the sham tDCS group, a return to baseline is expected in the follow-up measures.

Transcranial Direct Current Stimulation (tDCS): HDC stimulators (Newronika TM, Milan, Italy) will be used. For active stimulation, the current intensity will be constant at 2 mA, with a stimulation time of 20 minutes daily for 12 days, and an initial and final ramp of 30 seconds. For the placebo group, current will only be applied during the initial and final ramps to generate the sensation of active stimulation. A neoprene cap with carbon rubber electrodes and sponges soaked in saline solution (5 x 5 cm) will be used. The anode will be placed over the left dorsolateral prefrontal cortex (DLPFC), and the cathode over the right supraorbital area (rSO).

Cognitive Training (CT): The CT will consist of 12 sessions of 50 minutes each, based on tasks involving executive functions and memory, including categorization, answering questions, short stories, problem-solving, recalling autobiographical moments, planning simple tasks, and schedule analysis.

DETAILED DESCRIPTION:
As a preliminary step to this study, it should be noted that contact with patients will be obtained from the Neurology service at the Consorcio Hospital General Universitario. Before starting the research and to obtain subject participation, the service will inform potential participants about the possibility of being included in a study related to electrical stimulation, noting that they will have to receive intervention through transcranial Direct Current Stimulation (tDCS) and Cognitive Training (CT) for twelve days. Once an initial commitment to possible participation is obtained from the patients, they will be informed that they will receive a phone call from the research team at the University of Valencia to schedule an in-person appointment where they will be provided with detailed information.

During this first appointment, held at the assigned health center or specialty center, the intervention procedure will be explained in more detail, and informed consent will be obtained from those subjects who decide to participate. It is important to highlight that the information regarding the procedure will emphasize aspects related to the safety and tolerability of the treatment, adherence to it, and the ease of application given its home-based nature.

From this point, the clinical interview will aim to assess the general health status and assess compliance with inclusion and exclusion criteria.; a neuropsychological evaluation will also be performed, although participants will be given the option to undergo this first evaluation during a second appointment. It should be noted that the total duration of the evaluation for participants in the early dementia group may be approximately 50 minutes.

Once the baseline evaluation is available, a coordinated schedule with the participants will be set to establish the start of the treatment and its continuity for the assigned duration; this aspect is crucial as a commitment to continuity from the participants is necessary. To facilitate this, a flexible start date will be provided to avoid any planned interruptions during the process. Additionally, given its home-based nature, the necessary information for home visits will be obtained, and an approximate time for the intervention will be established to ensure consistency. For this process, a psychologist hired for this purpose will visit the homes of the participants to carry out the stimulation.

The main critical point of this project is believed to be treatment adherence. Multiple sessions require subjects to repeatedly travel to the treatment location, posing a significant and often insurmountable burden for patients and their caregivers, along with substantial time and cost for service providers, especially as sample size increases. This difficulty often results in a high dropout rate. Providing tDCS and CT treatment at home, as proposed in this project, can reduce the burden on patients and their families by eliminating the need to travel to medical or research facilities for each treatment session, promoting adherence and compliance with the treatment. Therefore, implementing the outlined procedure in this research appears necessary not only to evaluate clinical efficacy but also to ensure the correct execution of stimulations and prevent dropouts.

Additionally, it is believed that one of the strengths and a key contingency strategy for addressing the mentioned critical point is the team's ability to adapt to contact with this type of patient and their caregivers. In this regard, it is crucial to implement an innovative paradigm, already applied in previous projects and leading global healthcare transformation, known as Patient Centricity (patient-centered care). Patient participation and care are essential aspects of research and procedural development, as well as disease management. Health outcomes depend on patient involvement, and there is a clear need to partner with them in the research, development, implementation, and advancement of health procedures to achieve better results. Creating a patient-centered solution involves obtaining input from patients and their caregivers, as is the case with this project, and making decisions based on their needs and perspectives. Humanizing science contributes to better acceptance, improving patient relationships and safety, and helping to prevent errors.

Considering the study groups, 3 repeated measures (pre, post, and follow-up), a statistical power of 95%, and a 95% confidence interval with an estimated effect size of η² = 0.16, it is estimated that an N = 30 participants would be needed, which means 15 subjects per group. Additionally, two differentiated samples will be obtained to apply the intervention: patients with mild cognitive impairment and patients with early-stage Alzheimer's disease.

The data will be analyzed using mixed ANOVAs with 2 groups (active vs. sham; between subjects) x 3 evaluations (pre-intervention, post-intervention, and follow-up; within subjects). The efficacy of tDCS should be observed by finding a significant interaction between these two independent variables.

ELIGIBILITY:
Inclusion Criteria:

Prodromal Alzheimer's disease: score equal to or higher than 23 points on the MMSE and scores equal to level 3 on the Global Deterioration Scale (GDS).

Initial Alzheimer's disease: score equal to or higher than 18 points on the MMSE and scores equal to level 4 on the Global Deterioration Scale (GDS).

Exclusion Criteria:

subjects with contraindications to tDCS (metal implants, intracranial, intracranial hypertension), significant cerebrovascular disease or severe psychiatric symptoms.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Baseline to approximately 6 weeks
  The Mini-Mental State Examination (MMSE) was used as an index of global cognitive functioning; the maximum score is 30 points. This test was designed to estimate the existence and severity of cognitive impairment. Participants with scores equal to or below 23 will be considered cognitive deficient. Post-intervention minus baseline. Difference score range is (-30 to 30) with positive scores reflecting improvement.

SECONDARY OUTCOMES:
Direct and inverse digits of the Wechsler Intelligence Scale for Adults-III | Baseline to approximately 6 weeks
  Direct and inverse digits of the Wechsler Intelligence Scale for Adults-III assess attentional capacity by exposing the participant to increasing amounts of information. On the direct digits task, which is used to assess immediate recall, the subject must repeat the sequence of numbers in the same order in which they are read by the examiner. On the inverse digit task, which assesses working memory and mental flexibility, the subject must say the digits backwards from the way they were presented by the examiner. Both tests are evaluated in the same way, assigning one point for each correct item, with a maximum score of 16 for both tests. Post-intervention minus baseline. Difference score range is (-16 to 16) with positive scores reflecting improvement.
Complutense Verbal Learning Test (TAVEC) - Memory | Baseline to approximately 6 weeks
  The Complutense Verbal Learning Test (TAVEC) presents a list of 16 words that, after being read by the evaluator, have to be repeated by the participant. The list is repeated five times (trials); the participant is again asked to remember the 16 words. The test was administered to evaluate the participant's immediate memory (Trial 1), learning ability (Trial 5 ). Post-intervention minus baseline. Scale is scored 0-16. Difference score range is (-16 to 16) with positive scores reflecting improvement.

OTHER OUTCOMES:
Memory Alteration Test (M@T)- Cognitive Impairment | Baseline to approximately 6 weeks
  The Memory Alteration Test (M@T) provides efficient and valid screening for A-MCI and early-stage AD. The test evaluates different abilities such as: encoding, orientation, semantic memory, and free recall. The maximum score is 50 points. The optimal cut-off point for distinguishing mild cognitive impairment of the amnesiac type from subjective memory complaints is 37 points. The optimal cut-off point for Alzheimer's disease is 31 points. Post-intervention minus baseline. Scale is scored 0-50. Difference score range is (-50 to 50) with positive scores reflecting improvement.
Barcelona Test (BT) - Ability to Access and Recall Elements From the Lexical and Semantic Store | Baseline to approximately 6 weeks
  Barcelona Test (BT) assesses the ability to access and recall lexical and semantic items by means of 2 subtests: a. Semantic fluency: recall the highest number of words from the category 'animals' in one minute; b. Phonological fluency: recall the highest number of words beginning with the letter 'p' in three minutes. Minimum and maximum range for Semantic fluency and Phonological fluency: 0 to n (no upper limit). Method of calculation: Scores for each subtest are reported separately. No combined scores or averages between subtests are calculated. Interpretation: Good categorical recall is considered good when evoking more than 16 animals in 1 minute and good verbal fluency when evoking more than 19 words beginning with 'p' in 3 minutes. This test assesses the ability to access and recall items from the lexical and semantic store. Processes involved: processing speed, cognitive flexibility and working memory. Post-intervention less baseline with positive scores reflecting improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Melendez, PhD, Principal Investigator — University of Valencia
Locations (1):
- Universidad de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
The main reason for not sharing the individual participant data (IPD) description plan is to preserve the confidentiality and privacy of clinical trial participants. The protection of participants' personal and medical information is considered a top priority in this study.

REFERENCES:
- [Result] Melendez JC, Satorres E, Pitarque A, Delhom I, Real E, Escudero J. Effectiveness of tDCS at Improving Recognition and Reducing False Memories in Older Adults. Int J Environ Res Public Health. 2021 Feb 1;18(3):1317. doi: 10.3390/ijerph18031317. PMID 33535690
- [Result] Satorres E, Escudero Torrella J, Real E, Pitarque A, Delhom I, Melendez JC. Home-based transcranial direct current stimulation in mild neurocognitive disorder due to possible Alzheimer's disease. A randomised, single-blind, controlled-placebo study. Front Psychol. 2023 Jan 3;13:1071737. doi: 10.3389/fpsyg.2022.1071737. eCollection 2022. PMID 36660288
- [Result] Satorres E, Melendez JC, Pitarque A, Real E, Abella M, Escudero J. Enhancing Immediate Memory, Potential Learning, and Working Memory with Transcranial Direct Current Stimulation in Healthy Older Adults. Int J Environ Res Public Health. 2022 Oct 5;19(19):12716. doi: 10.3390/ijerph191912716. PMID 36232016
- [Result] Hill AT, Fitzgerald PB, Hoy KE. Effects of Anodal Transcranial Direct Current Stimulation on Working Memory: A Systematic Review and Meta-Analysis of Findings From Healthy and Neuropsychiatric Populations. Brain Stimul. 2016 Mar-Apr;9(2):197-208. doi: 10.1016/j.brs.2015.10.006. Epub 2015 Oct 23. PMID 26597929
- [Result] Bahar-Fuchs A, Martyr A, Goh AM, Sabates J, Clare L. Cognitive training for people with mild to moderate dementia. Cochrane Database Syst Rev. 2019 Mar 25;3(3):CD013069. doi: 10.1002/14651858.CD013069.pub2. PMID 30909318
- [Result] Gates NJ, Vernooij RW, Di Nisio M, Karim S, March E, Martinez G, Rutjes AW. Computerised cognitive training for preventing dementia in people with mild cognitive impairment. Cochrane Database Syst Rev. 2019 Mar 13;3(3):CD012279. doi: 10.1002/14651858.CD012279.pub2. PMID 30864747